CLINICAL TRIAL: NCT01505842
Title: Randomized Controlled Trial (RCT) to Compare Dysplasia Detection Rate in Colonoscopy Without Chromoendoscopy Versus Colonoscopy With Chromoendoscopy in Detecting Dysplasia in Ulcerative Colitis and Crohn's Colitis Patients.
Brief Title: Chromoendoscopy for Dysplasia Detection in Chronic Inflammatory Bowel Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Peter Thelin Schmidt, Head of Endoscopy, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PTS-01
Record Dates: First submitted 2011-12-29; First posted 2012-01-09 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Ulcerative Colitis; Crohn's Colitis
Keywords: Ulcerative colitis; Crohn's disease; Chromoendoscopy; Dysplasia; Neoplasia; Inflammatory Bowel Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease; Neoplasms; Inflammatory Bowel Diseases | interventions — Colonoscopy; Indigo Carmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Colonoscopy with chromoendoscopy (Experimental): Colonoscopy with chromoendoscopy using 0.2-0.5% Indigo-Carmine solution sprayed in the whole colon and rectum plus 32 random biopsies plus biopsies from suspicious areas
  Interventions: Procedure: Colonoscopy with Indigo-Carmine chromoendoscopy
- Conventional colonoscopy (Active Comparator): White light colonoscopy plus 32 random biopsies plus biopsies from suspicious areas
  Interventions: Procedure: Conventional white-light colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy with Indigo-Carmine chromoendoscopy — Colonoscopy with chromoendoscopy using 0.2-0.5% Indigo-Carmine solution sprayed in the whole colon and rectum plus 32 random biopsies plus biopsies from suspicious areas
  Other Names: Indigo-Carmine
  Arms: Colonoscopy with chromoendoscopy
Procedure: Conventional white-light colonoscopy — White light colonoscopy plus 32 random biopsies plus biopsies from suspicious areas
  Arms: Conventional colonoscopy

SUMMARY:
Patients with longstanding ulcerative colitis or crohn's disease in the large bowel have an increased risk of developing cancer. The purpose of this study is to determine if visualizing of the mucosa in details using a dye spray (indigo-carmine) will result in detection of more abnormalities than conventional colonoscopy without dye spray.

DETAILED DESCRIPTION:
Background: Patients with ulcerative colitis and Crohn's colitis are at increased risk of colon cancer. The usefulness of chromoendoscopy is debated. Previous studies are either based on magnifying endoscopy or on non-randomized trials. Some guidelines recommend chromoendoscopy with targeted biopsies and some normal colonoscopy with up to 40 random biopsies.

Chromoendoscopy has the ability to identify subtle lesions that are otherwise missed by standard endoscopy. Whether chromoendoscopy with targeted biopsies can replace standard colonoscopy with random biopsies in the surveillance of patients with chronic colitis is unknown.

Aim: In a RCT in surveillance colonoscopies in patients with ulcerative colitis or Crohn's colitis, we will determine if chromoendoscopy using a dilute solution of Indigo-carmine will improve dysplasia detection rate compared with colonoscopy without chromoendoscopy.

Methods: After informed consent patients undergoing surveillance colonoscopy will be randomized to be examined by the study or control method. The study method will employ a 0.2-0.5% Indigo-Carmine solution sprayed over the colonic and rectal mucosa. The control method will be colonoscopy without Indigo-Carmine chromoendoscopy. In both the study arm and the control arm all subjects will have 32 random biopsies taken (4 from each of 8 defined segments of the colon) and biopsies from suspicious mucosa.

ELIGIBILITY:
Inclusion Criteria:

Patients with ulcerative colitis or Crohn's colitis satisfying criteria for surveillance colonoscopy:

* Ulcerative colitis, extensive > 8 years OR Crohn's colitis involving ≥ 1/3 of colon/rectum
* history of PSC or
* history of previous dysplasia on colon biopsies or
* family history of colon cancer in first degree relative

Exclusion Criteria:

* Patients who decline to participate
* Unable to give informed consent
* Increased risk of bleeding (i.e. Warfarin, bleeding disorders, Clopidogrel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2011-02; Primary Completion 2019-04-04 (Estimated); Study Completion 2019-04-04 (Estimated)

PRIMARY OUTCOMES:
Prevalence of dysplastic lesions | 12 month
  Number of patients with dysplastic lesions by colonoscopy with chromoendoscopy using Indigo-carmine versus colonoscopy without chromoendoscopy

SECONDARY OUTCOMES:
Number and rate of targeted and non-targeted biopsies detecting dysplasia and non-dysplasia | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Peter T Schmidt, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karoliniska University Hospital, Dept. of Gastroenterology, Stockholm, Sweden

REFERENCES:
- [Derived] Alexandersson B, Hamad Y, Andreasson A, Rubio CA, Ando Y, Tanaka K, Ichiya T, Rezaie R, Schmidt PT. High-Definition Chromoendoscopy Superior to High-Definition White-Light Endoscopy in Surveillance of Inflammatory Bowel Diseases in a Randomized Trial. Clin Gastroenterol Hepatol. 2020 Aug;18(9):2101-2107. doi: 10.1016/j.cgh.2020.04.049. Epub 2020 Apr 27. PMID 32353535